CLINICAL TRIAL: NCT02949401
Title: Stress Inoculation Through Virtual Reality in the Pediatric Electrophysiology Laboratory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anne M. Dubin, Professor of Pediatrics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 37603
Record Dates: First submitted 2016-10-19; First posted 2016-10-31 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Stress, Psychological; Stress, Physiological; Anxiety; Pain Perception
Keywords: Virtual Reality; Stress Inoculation; Procedure
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): No research intervention to be administered.
  Participants will have standard preparation for a procedure including discussion of the procedure with the provider the day before the procedure with all questions answered at that time.
- Virtual Reality (Experimental): The VR interactive module will consist of a 360° visit to the Hospital where patients encounter the various aspects of a procedure from the front door; through the pre-operative area where patients will receive an IV; to the catheterization lab and placement of the anesthesia mask; and back to the post anesthesia care unit. Patients will be accompanied by a child who acts as a guide to the experience. The guide will help explain what the patient is seeing and what to expect along the way. Health care professionals will be enmeshed within the scenarios and will also help with the explanations along the way. Patients will be prompted to enter the relaxation scenarios at different stressful times along the tour to practice relaxation and mindfulness techniques (i.e. before IV start, or upon entering catheterization laboratory). Relaxation scenarios will include a snow scene, tropical beach or other guided imagery scenes.
  Interventions: Behavioral: Use of Virtual Reality App

INTERVENTIONS:
Behavioral: Use of Virtual Reality App — The VR app will consist of relaxation techniques as well as a virtual tour of the hospital (pre-op area, IV placement, cath lab, and post-op area).
  Arms: Virtual Reality

SUMMARY:
The goal of this study is to assess the utility of virtual reality technology to aid in the mental health of patients with cardiac disease, specifically looking at decreasing anxiety and perceptions of pain from stressful procedures in the pediatric electrophysiology laboratory.

DETAILED DESCRIPTION:
The investigators will perform a pilot study of 40 patients who are randomized to either standard of care preparation for an electrophysiology procedure (control arm) vs. Virtual Reality preparation (VR arm). Participants in control arm will have standard preparation for a procedure including discussion of the procedure with the provider the day before the procedure with all questions answered at that time. VR arm participants will have access to the Virtual Reality tour and gear 1 week prior to the procedure. VR arm participants will be instructed to watch the Virtual Reality tour at least three times prior to the procedure but will be encouraged to watch as often as the participants would like. The Virtual Reality equipment will measure how often participants complete the tour. All participants will undergo anxiety measures a total of four times: once at time of recruitment, day of procedure and then 1 week and 4 weeks post procedure. Participants will have cortisol salivary swabs performed 1 week before procedure (before VR use), pre-op visit, day of procedure, and immediately following procedure. Heart rate and blood pressure will be measured on day of procedure.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric Cardiology patients between the age of 10 and 20 years old
* Undergoing cardiac electrophysiology procedure

Exclusion Criteria:

* Inability to wear virtual reality glasses
* Patients under 10 years old
* Prior psychiatric illness

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
Change in anxiety levels from baseline in patients as measured by the State Trait Anxiety Inventory (STAI). | At time of recruitment, day of procedure, 1 week post procedure, and 4 weeks post procedure
  State -Trait Anxiety Inventory (STAI) is a widely used self-report measure that estimates situational (state) and baseline (trait) anxiety in adults and children. It is both valid and reliable and routinely used in measuring anxiety associated with medical procedures. The pediatric version is available for use with upper elementary, or junior high or high school aged children.

SECONDARY OUTCOMES:
Change in anxiety levels from baseline in patients as measured by Visual Analog Scale of Anxiety | At time of recruitment, day of procedure
  Visual Analog Scale of Anxiety (VAS) is a widely used self-reported and observational measure of anxiety. Patients place a vertical line along a 10 cm horizontal line which is anchored with the descriptors "not at all anxious" and "extremely anxious" and 10 markings 1 cm apart. This simple format of assessing anxiety is often used in operating rooms or before medical procedures given its brevity and ease of administration is fast-paced settings. It has been correlated with STAI scores.
Change in parent observation of child behavior from baseline as measured by Child Behavior Checklist (CBCL) | At time of recruitment and 4 weeks post procedure
  Child Behavior Checklist (CBCL) is a rating form of child behavior completed by parents. It has been developed for children aged 6-18 years. This checklist groups into sets of behaviors: internalizing, externalizing and total problems.
Change in anxiety levels from baseline in parents as measured by parental STAI | At time of recruitment, day of procedure, 1 week post procedure, and 4 weeks post procedure
  State -Trait Anxiety Inventory (STAI) is a widely used self-report measure that estimates situational (state) and baseline (trait) anxiety in adults and children. It is both valid and reliable and routinely used in measuring anxiety associated with medical procedures.
Change in salivary cortisol levels from baseline in patients | 1 week before procedure (before use of VR), Day of pre-op, Day of procedure, Day after procedure or immediately after procedure if outpatient
Heart rate in patients | Day of procedure
blood pressure in patients | Day of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Anne Dubin, MD, Principal Investigator — Stanford University; Lauren Schneider, PsyD, Principal Investigator — Stanford University; Danton Char, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University / Lucile Packard Children's Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kain ZN, Caramico LA, Mayes LC, Genevro JL, Bornstein MH, Hofstadter MB. Preoperative preparation programs in children: a comparative examination. Anesth Analg. 1998 Dec;87(6):1249-55. doi: 10.1097/00000539-199812000-00007. PMID 9842807
- [Background] Kain ZN, Mayes LC, O'Connor TZ, Cicchetti DV. Preoperative anxiety in children. Predictors and outcomes. Arch Pediatr Adolesc Med. 1996 Dec;150(12):1238-45. doi: 10.1001/archpedi.1996.02170370016002. PMID 8953995
- [Background] Pallavicini F, Gaggioli A, Raspelli S, Cipresso P, Serino S, Vigna C, Grassi A, Morganti L, Baruffi M, Wiederhold B, Riva G. Interreality for the management and training of psychological stress: study protocol for a randomized controlled trial. Trials. 2013 Jun 28;14:191. doi: 10.1186/1745-6215-14-191. PMID 23806013
- [Background] Gold JI, Kim SH, Kant AJ, Joseph MH, Rizzo AS. Effectiveness of virtual reality for pediatric pain distraction during i.v. placement. Cyberpsychol Behav. 2006 Apr;9(2):207-12. doi: 10.1089/cpb.2006.9.207. PMID 16640481
- [Background] Sander Wint S, Eshelman D, Steele J, Guzzetta CE. Effects of distraction using virtual reality glasses during lumbar punctures in adolescents with cancer. Oncol Nurs Forum. 2002 Jan-Feb;29(1):E8-E15. doi: 10.1188/02.ONF.E8-E15. PMID 11845217
- [Background] Fortier MA, Del Rosario AM, Martin SR, Kain ZN. Perioperative anxiety in children. Paediatr Anaesth. 2010 Apr;20(4):318-22. doi: 10.1111/j.1460-9592.2010.03263.x. Epub 2010 Feb 23. PMID 20199609
- [Background] Folstein MF, Luria R. Reliability, validity, and clinical application of the Visual Analogue Mood Scale. Psychol Med. 1973 Nov;3(4):479-86. doi: 10.1017/s0033291700054283. No abstract available. PMID 4762224
- [Background] Davey HM, Barratt AL, Butow PN, Deeks JJ. A one-item question with a Likert or Visual Analog Scale adequately measured current anxiety. J Clin Epidemiol. 2007 Apr;60(4):356-60. doi: 10.1016/j.jclinepi.2006.07.015. Epub 2006 Dec 27. PMID 17346609
- [Background] Tunc-Tuna P, Acikgoz A. The Effect of Preintervention Preparation on Pain and Anxiety Related to Peripheral Cannulation Procedures in Children. Pain Manag Nurs. 2015 Dec;16(6):846-54. doi: 10.1016/j.pmn.2015.06.006. Epub 2015 Aug 17. PMID 26293196